CLINICAL TRIAL: NCT02478892
Title: Preliminary Evaluation of Screening for Pancreatic Cancer in Patients With Inherited Genetic Risk
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 26214
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: high risk; specifically those with BRCA1/2 mutations
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Up to 40mL of blood may be collected for analysis at each screening examination.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Collection of data from endoscopic ultrasound or MRI/MRCP of the abdomen — Participants in this study should be undergoing pancreatic cancer screening with endoscopic ultrasound or MRI as part of their standard care. These should typically be done at least every 12 months, and the imaging tests will be ordered as routine clinical tests and will be billed to the participant's insurance. This study does not cover the costs of these screening tests, however the study will track the results of these screening tests.
Other: Blood sample collection for research — Up to 40mL of blood may be collected for analysis at each screening examination.

SUMMARY:
The study is a prospective, observational study evaluating the utility of endoscopic ultrasound or MRI for the identification of preneoplastic and neoplastic pancreatic lesions in patients at high risk for pancreatic cancer, specifically those with BRCA1/2, ATM, or PALB2 mutations.

DETAILED DESCRIPTION:
Endoscopic Ultrasound (EUS) has emerged as a critical component in the imaging, staging, and diagnosis of pancreatic cancer. Not only can EUS delineate a mass utilizing sonography through the wall of the stomach or duodenum, but it also can obtain diagnostic fine needle aspiration of suspicious lesions. Especially in patients with incomplete visualization of a mass on cross-sectional imaging, EUS can provide valuable anatomic information prior to surgical exploration. While several studies have demonstrated that EUS has high sensitivity and specificity in diagnosing pancreatic masses, head-to-head comparisons with established modalities like CT have been often methodologically flawed. In a meta-analysis, it was found that of 4 studies that assessed resectability, 2 showed no difference and 1 favored each modality. As such, estimates of accuracy for assessing preoperative resectability have also ranged in several studies from 63-93%. As such it has been recognized as an accepted modality for the evaluation of potential pancreatic malignancy.

While pancreatic ductal adenocarincoma (PDAC) screening in the general population is not feasible given the low incidence of PDAC, screening in high risk cohorts may allow for early detection of resectable, and potentially curable tumors. Clinical outcome of patients with smaller, non-metastasized tumors have a significantly improved 5-year survival. Generally the current recommendation is that patients who are first degree relatives of patients with PDAC from a familial PDAC kindred with at least 2 directly related relatives, patients with Peutz-Jeghers syndrome, those with a CDKN2A pathogenic germline variant, and those with BRCA1/BRCA2/ATM/PALB2/Lynch pathogenic germline variants with a first or second degree relative with pancreatic cancer would qualify for pancreatic cancer screening. However, there is continued debate about whether family history should be used to determine who is eligible for pancreatic cancer screening. In this study we will be following individuals at the University of Pennsylvania who have a BRCA1, BRCA2, ATM, or PALB2 pathogenic germline variant and who are getting pancreatic cancer screening, regardless of whether or not they have a family history of PDAC. Ultimately, in high-risk individuals, such as BRCA1/2, ATM, and PALB2 carriers, the successful identification of early neoplastic/preneoplastic lesions of the pancreas would allow for timely intervention and likely improved survival in this cohort.

ELIGIBILITY:
Inclusion Criteria

* Age >= 18
* Documented germline pathogenic or likely pathogenic BRCA1, BRCA2, ATM, or PALB2 mutation
* If no history of PDAC in a first or second degree relative, age >= 50
* If there is a history of PDAC in a first or second degree relative, minimum age of eligibility is 10 years younger than the age of onset of the youngest relative with pancreatic cancer

Exclusion Criteria

• Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk for pancreatic cancer, specifically those with pathogenic germline variant in BRCA1, BRCA2, ATM, or PALB2 who will be undergoing pancreatic cancer screening as part of their routine clinical care.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
identifying pancreatic neoplastic lesions lesions in patients with BRCA1/2 mutations and other less common, but related mutations (ATM, PALB2) as well as mutations identified in the future. | 10 years
  The primary objective of the study is the observational screening of patients with BRCA1/2, ATM, or, PALB2 mutations for pancreatic neoplastic lesions, to assess for both the feasibility of this approach in this high risk population as well as to better establish the incidence of these lesions in this cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Katona BW, Long JM, Ahmad NA, Attalla S, Bradbury AR, Carpenter EL, Clark DF, Constantino G, Das KK, Domchek SM, Dudzik C, Ebrahimzadeh J, Ginsberg GG, Heiman J, Kochman ML, Maxwell KN, McKenna DB, Powers J, Shah PD, Wangensteen KJ, Rustgi AK. EUS-based Pancreatic Cancer Surveillance in BRCA1/BRCA2/PALB2/ATM Carriers Without a Family History of Pancreatic Cancer. Cancer Prev Res (Phila). 2021 Nov;14(11):1033-1040. doi: 10.1158/1940-6207.CAPR-21-0161. Epub 2021 Aug 2. PMID 34341011